CLINICAL TRIAL: NCT02004405
Title: The Study of Heart Rate Variability in Patients With Fibromyalgia - Effects of Strengthening Exercises
Brief Title: Heart Rate Variability in Fibromyalgia - Effects of Strengthening Exercises
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Espirito Santo (Other)
Responsible Party: Principal Investigator, Valéria Valim, PhD, MD Valéria Valim, Federal University of Espirito Santo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUES01
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Fibromyalgia
Keywords: autonomic nervous system; fibromyalgia; autonomic dysfunction; strengthening; flexibility; exercise; heart rate variability
MeSH Terms: conditions — Fibromyalgia; Primary Dysautonomias; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- strengthening exercise (Experimental): The experimental group (STRE) will receive strengthening training in "Station for lifting weight exercises" (Flex Mega 8, Flex Fitness Equipment Brand) using the recommendations of the American College of Sports Medicine (ACMS, 2010), twice a week, during 45 minutes for 16 weeks.
  Interventions: Other: strengthening exercise
- Flexibility exercise (Active Comparator): The control group (FLEX) will receive stretching and flexibility exercise training according to the protocol of prescription and previously tested and described in appendix F (Valim et al., 2003), twice a week, during 45 minutes for 16 weeks.
  Interventions: Other: flexibility exercise

INTERVENTIONS:
Other: strengthening exercise — The experimental group (STRE) will receive strengthening training in "Station for lifting weight exercises" (Flex Mega 8, Flex Fitness Equipment Brand) using the recommendations of the American College of Sports Medicine (ACMS, 2010), twice a week, during 45 minutes for 16 weeks.
  Arms: strengthening exercise
Other: flexibility exercise — The control group (FLEX) will receive stretching and flexibility exercise training according to the protocol of prescription and previously tested and described in appendix F (Valim et al., 2003), twice a week, during 45 minutes for 16 weeks.
  Arms: Flexibility exercise

SUMMARY:
Abstract Objective: Autonomic dysfunction is an important mechanism that could explain many symptoms observed in fibromyalgia (FM). Exercise is an effective treatment, with benefits potentially mediated through changes in autonomic modulation. Strengthening is one of the less studied exercises in FM, and the acute and chronic effects of strengthening on the autonomic system remain unknown. The objective of this study is to assess the effects of strengthening exercises (STRE) on autonomic modulation, pain perception and the quality of life (QOL) of FM patients. Methods: Sedentary women with FM (ACR 1990) will be randomly selected to STRE or flexibility (FLEX) exercises in a blind controlled trial. The intensity of STRE will be set at 45% of the estimated load of 1 Repetition Maximum (RM) in 12 different exercises. The primary outcomes will be pain measured using the Visual Analog Scale (VAS) and the Heart Rate Variability (HRV) analysis. Other outcomes will be assess: fitness measured by treadmill test, the sit and reach test (Wells and Dillon's Bench), handgrip dynamometry; and quality of life by the Fibromyalgia Impact Questionnaire (FIQ), the Beck and Idate Trait-State Inventory (IDATE), a short-form health survey (SF-36). Statistical analyses and ethical procedures: The visual analog scale (VAS) for pain will be the primary measure used to determine sample size. Statistical significance will be set at 5% and power of 80%. These led to at least 58 participants to be randomized. The main hypothesis is that strengthening exercise is a better treatment than flexibility exercise to improve pain, HRV and quality of life. In all measures tested we will consider the null hypothesis (H0) as being the point of equality between groups tested and H1 the point of difference. Bilateral tests were carried out adopting a 5% level of significance. The normality of the results will be tested using the Shapiro-Wilk test. Student's "t"-test for paired samples will be used to perform intra-group comparisons at different times, when the data were normally distributed, and the nonparametric equivalent of Student's t-test (Wilcoxon test) will be used when the data show an asymmetrical distribution. To compare the data between the STRE and FLEX groups, ANOVA for repeated measures will be used, followed by post-hoc Bonferroni's test.

DETAILED DESCRIPTION:
STUDY PROTOCOL: The experimental group (STRE) will receive strengthening training in "Station for lifting weight exercises" (Flex Mega 8, Flex Fitness Equipment Brand) using the recommendations of the American College of Sports Medicine (ACMS, 2010), twice a week, during 45 minutes for 16 weeks. The control group (FLEX) will receive stretching and flexibility exercise training according to the protocol of prescription and previously tested and described in appendix F (Valim et al., 2003), twice a week, during 45 minutes for 16 weeks. The minimum number of patients per group will be 30. The randomization will be by arriving order of the patients at the Clinic, having 2 groups with a distribution at random one by one. There will be an examiner for the selection and unblinded randomization and another for the application of tools that will be blind. Patients will undergo clinical and cardiological evaluation with an exercise stress test (Ergometric test) request in all of them according to ACMS as one more method of evaluation for inclusion and exclusion.

The evaluation will be performed by a blind examiner, an expert physiotherapist in rheumatology and trained for the application of the tools at the beginning, after 30, 60, 90, 120 days from the treatment onset.

The measure for prescription and muscle strength gain will be by the method of maximal repetitions (Lindh et al., 1994; Tritschler, 2003; Brosseau et al., 2008; ACSM, 2010). The evaluations will take place at the beginning, 30, 60, 90, 120 days (final evaluation). Evaluations will be performed by the same blind examiner for the examined group. The training team will be formed by a physiotherapist, physical educator, and experienced doctors at strengthening training and flexibility and stretching exercises and they must follow the following protocol.

PROTOCOL OF EXERCISES The strength training will be performed according to American College of Sports Medicine (ACSM) and will have a mild to moderate intensity representing 45% of the estimated 1RM obtained from the maximal repetition method. Eight major muscle groups will be trained (quadriceps femoris, hamstrings, biceps brachii, triceps brachii, pectoral, calf, deltoid, and latissimus dorsi) in 12 different exercises, with 3 sets of 12 repetitions (leg Press, leg extension, hip flexion, pectoral fly, triceps extension, shoulder flexion, leg curl, calf, pulldown, shoulder abduction, biceps flexion and shoulder extension). Theses 12 different exercises will be distributed in a composed circuit system of 2 sets of exercises: Set A ((leg Press, leg extension, hip flexion, pectoral fly, triceps extension, shoulder flexion) and set B (leg curl, calf, pulldown, shoulder abduction, biceps flexion and shoulder extension). Each set will be applied once a week alternatively. The exercises will be performed twice a week during 16 weeks.

During the training process a load increase will be performed in order to seek progressive muscle strengthening improvement in a controlled way and according to patients' clinical evolution. Blood pressure and heart rate will be monitored as well.

Strength and strengthening training will be performed at the Evaluation, Physical Conditioning and Rehabilitation Laboratory (LACORE) at the University Hospital in in Federal University of Espirito Santo.

We have chosen the frequency of twice a week because it is a frequency (for this kind of study) validated in the literature (Figueroa et al., 2008, Kingsley et al., 2009; 2010).

ELIGIBILITY:
Inclusion Criteria:

* Classification criteria for Fibromyalgia (ACR 1990)
* Sedentary subjects (without regular physical activity in the last 3 months)
* Women between 18 to 65 years old

Exclusion Criteria:

* Cardiovascular and/or respiratory diseases that might limit physical activity (COPD, Pulmonary Fibrosis, asthma moderate to severe, respiratory insufficiency);
* Organ dysfunction (renal, hepatic, coronary, pulmonary insufficiency);
* Arterial hypertension and diabetes mellitus;
* Uncontrolled thyroid disease;
* Autoimmune rheumatic diseases and/or non-autoimmune with symptoms that might limit the movement or physical effort;
* The use of beta blockers, calcium channel blockers and any other anti-hypertensive, anticonvulsants; non tricycles antidepressants; opioid analgesic including tramadol.
* cyclobenzaprine >10 mg/day, and amtriptyline > 25 mg/day;
* Performing or have performed exercise within the last 3 months;
* Inability to understand the questionnaires;
* Positive treadmill test for myocardial ischemia;
* Receipt of the social security benefits.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
pain | 4 weeks
  Visual analogic scale

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire | Initial, 8 weeks, 16 weeks
  Symptoms
Short Form Health Survey | Initial, 8 weeks, 16 weeks
State-Trait Anxiety Inventory (IDATE) | initial, 8 weeks, 16 weeks
  Mood evaluation
BECK Depression Inventory | Initial, 8 weeks, 16 weeks
  Mood evaluation
Treadmill test | initial and 16 weeks
  cardiorespiratory fitness cardiovascular risk
Sit and Reach Test | 4 weeks
  flexibility
dynamometry | 4 weeks
  global strength
Maximal repetition test | 4 weeks
  muscle strength
autonomic modulation | 4 weeks
  Ratio low frequecy to high frequency in the Heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bernadete RO Gavi, Master, Principal Investigator — Federal University of Espírito Santo
Locations (1):
- Valéria Valim, Vitória, Espírito Santo, Brazil

REFERENCES:
- [Derived] Gavi MB, Vassalo DV, Amaral FT, Macedo DC, Gava PL, Dantas EM, Valim V. Strengthening exercises improve symptoms and quality of life but do not change autonomic modulation in fibromyalgia: a randomized clinical trial. PLoS One. 2014 Mar 20;9(3):e90767. doi: 10.1371/journal.pone.0090767. eCollection 2014. PMID 24651512